CLINICAL TRIAL: NCT04098211
Title: Longitudinal Assessment of Atypical Tripeptidyl Peptidase 1 Enzyme Deficiency (Neuronal Ceroid Lipofuscinosis Type 2) Patients
Brief Title: Longitudinal Assessment of Atypical Tripeptidyl Peptidase 1 Enzyme Deficiency Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Sponsor
Other Study IDs: 190219
Record Dates: First submitted 2019-07-22; First posted 2019-09-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Neuronal Ceroid-Lipofuscinoses; Neuronal Ceroid Lipofuscinosis CLN2; Spinocerebellar Ataxia, Autosomal Recessive 7
Keywords: Neuronal Ceroid Lipofuscinosis; Atypical CLN2 Disease; Natural History
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses; Spinocerebellar Ataxia, Autosomal Recessive 7

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to gather information on the possible symptoms that patients with atypical neuronal ceroid lipofuscinosis type 2 (also known as aTPP1 or atypical tripeptidyl peptidase deficiency) have and how they change over time.

DETAILED DESCRIPTION:
This study aims characterize the natural history of atypical TPP1 deficiency patients via longitudinal multidisciplinary assessments.

Multifaceted clinical, laboratory, imaging, and diagnostic assessments will be performed at regular intervals upon enrolled aTPP1 deficiency patients, collated, and analyzed over a three-year longitudinal period.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with documented TPP1 enzymatic deficiency or TPP1 sequence variants
* Onset of first symptom after 4 years of age
* Parental provision of informed consent; child provision of assent (if necessary)

Exclusion Criteria:

* Any patient with "Classical" TPP1 deficiency (onset of first symptom prior to 4 years of age)
* Investigator assessment that patient is not suitable candidate to participate in the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with documented TPP1 enzymatic deficiency or TPP1 sequence variants with onset of first symptom after 4 years of age
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
CLN2 Disease Severity Scoring | At baseline and every 3 months afterwards, up to 3 years
  Modified Hamburg Rating Scale. The rating scale consists of two domains (motor function, language). Within each domain, a score from 0 to 3 is assigned and overall scores are calculated by summing the domain scores for final rating of 0 (severely impaired) to 6 (normal).
Electroretinogram (ERG) | At baseline and every 6 months afterwards, up to 3 years
  Standard ERG will be performed to measure function of cones and rods of the inner and outer photoreceptor layers which amplitudes are typically decreased in classical TPP1 deficiency.
Optical Coherence Tomography (OCT) | At baseline and every 6 months afterwards, up to 3 years
  OCT is non-invasive, quantitative measurement of inner and outer photoreceptor layer thicknesses.
Gait Assessment | At baseline and every 6 months afterwards, up to 3 years
  Gait assessment is acquired utilizing infrared sensors applied to participant's clothing and will include collection of walking speed, cadence, swing phase, stride length and time, walking base width, stance phase, and double limb support phase.
Brain Magnetic Resonance Imaging (MRI) | At baseline and every 12 months afterwards, up to 3 years
  Pre/post-contrast images will be acquired to perform volumetric studies and white matter assessment.
Electroencephalography (EEG) | At baseline and every 12 months afterwards, up to 3 years
  EEG will be obtained and analyzed for changes that may be distinctive for TPP1 deficiency. Evaluation of background activity, mild/moderate/severe slowing for age.
Electroencephalography (EEG) | At baseline and every 12 months afterwards, up to 3 years
  EEG will be obtained and analyzed for changes that may be distinctive for TPP1 deficiency. Interictal discharges: location, focal/generalized, discharge burden.
Electroencephalography (EEG) | At baseline and every 12 months afterwards, up to 3 years
  Seizures.
Electroencephalography (EEG) | At baseline and every 12 months afterwards, up to 3 years
  Photoparoxysmal response: present/absent
Cognitive Assessment, Wechsler Intelligence Scale for Children version 4 (WISC-IV) | At baseline and every 12 months afterwards, up to 3 years
  WISC-IV will generate a full scale of intelligence quotient and five primary index scores: Verbal Comprehension, Visual Spatial, Fluid Reasoning, Working Memory, and Processing Speed. The WAIS-IV is scored by summing the raw scores for each subtest; each raw subtest score is then converted to a scaled scored. They are then combined to create a Full Scale IQ Index score. Test takers will also be given a score on the General Ability Index (GAI).
CSF Testing | At baseline and every 3 months afterwards, up to 3 years
  Standard laboratory testing and biobanking / storage of remaining CSF (via Ommaya if on enzyme replacement; via lumbar puncture if not on enzyme replacement)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States